CLINICAL TRIAL: NCT06331143
Title: Comparison of Analgesic Efficacy of Mid-Transverse Process to Pleura (MTP) Block and Intrathecal Morphine in Idiopathic Scoliosis Patients Undergoing Posterior Spinal Fusion: A Randomized Clinical Trial
Brief Title: Analgesic Efficacy of Mid-Transverse Process to Pleura (MTP) Block and Intrathecal Morphine in Idiopathic Scoliosis Patients Undergoing Posterior Spinal Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR551/2/24
Record Dates: First submitted 2024-03-17; First posted 2024-03-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Mid-Transverse Process Block; Intrathecal Morphine; Idiopathic Scoliosis; Posterior Spinal Fusion
MeSH Terms: interventions — Dental Occlusion; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mid-Transverse Process block (MTP) group (Experimental): Patients will receive mid-transverse process to pleura (MTP) block after induction of anesthesia.
  Interventions: Device: Ultrasound-Guided Mid-Transverse Process to Pleura (MTP) Block
- Intrathecal morphine (IM) group (Experimental): Patients will receive intrathecal morphine in a dose of 12 μg/kg (max 1000 μg) immediately after induction of anesthesia.
  Interventions: Drug: Morphine

INTERVENTIONS:
Device: Ultrasound-Guided Mid-Transverse Process to Pleura (MTP) Block — Patients will receive MTP block after induction of anesthesia.
  Arms: Mid-Transverse Process block (MTP) group
Drug: Morphine — Patients will receive intrathecal morphine in a dose of 12 μg/kg (max 1000 μg) immediately after induction of anesthesia.
  Arms: Intrathecal morphine (IM) group

SUMMARY:
The aim of this study is to compare the analgesic efficacy of mid-transverse process to pleura (MTP) block and intrathecal morphine in idiopathic scoliosis patients undergoing posterior spinal fusion surgery.

DETAILED DESCRIPTION:
The postoperative period for idiopathic scoliosis patients undergoing posterior spinal fusion (PSF) is fraught with challenges, including adequate postoperative pain control and prolonged hospitalization.

Intrathecal opioids have been used to manage postoperative pain in pediatric patients for a wide variety of surgeries , including adolescent and adult PSF. Multimodal analgesic (MMA) regimens using several drugs and techniques are considered to be necessary for postoperative pain relief.

The mid-transverse process to pleura (MTP) block was first described as a modified paravertebral block in 2017. The local anesthetics (LAs) are administered between the transverse process and the pleura. This results in a LA spread to the dorsal and ventral rami in the paravertebral space through the fenestrations in the superior costotransverse ligament at the level of injection, and frequently to adjacent levels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Idiopathic scoliosis patients undergoing posterior spinal fusion surgery.

Exclusion Criteria:

* Patient with morbid obesity (body mass index >40 kg/m2).
* Patients with pre-existing infection at block site.
* Known allergy to study drugs.
* Coagulation disorder.
* History of psychiatric illness.
* Pre-existing neurological deficits.
* Presence of any pre-operative pain or history of chronic pain.
* History of regular analgesic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-01-04 (Actual); Study Completion 2026-01-04 (Actual)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperative
  Degree of pain will be assessed by the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
  It will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.

SECONDARY OUTCOMES:
Heart rate | Till the end of surgery.
  Heart rate will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Mean arterial pressure | Till the end of surgery.
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Patient satisfaction | 24 hours postoperative.
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
  It will be assessed 24 hours after surgery.
Complications | 24 hours postoperative.
  Complications such as bradycardia, hypotension, nausea, vomiting, Pruritis, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S ElSharkawy, MD, Principal Investigator — Faculty of Medicine, Tanta University, Tanta, Egypt.
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author